CLINICAL TRIAL: NCT04297735
Title: Telemedicine Enabling Patients in Self-care Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Kathleen Fasing, Nurse Practioner, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00156966
Record Dates: First submitted 2020-02-28; First posted 2020-03-05 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Arrythmia
Keywords: telemedicine; self-care
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care group (Active Comparator): Discuss new arrhythmias, review symptoms, discuss methods to help symptoms, questions and answers, monitor devices every 3 months
  Interventions: Other: Standard of care group
- Telemedicine group (Experimental): Discuss new arrhythmias, review symptoms, discuss methods to help symptoms, questions and answers, monitor devices every 3 months
  Interventions: Behavioral: Telemedicine group; Behavioral: Telemedicine

INTERVENTIONS:
Other: Standard of care group — Visits every 6 months is standard of care.
  Other Names: Telemedicine
  Arms: Standard of care group
Behavioral: Telemedicine group — Conduct monthly telemedicine 'skype' visit
  Arms: Telemedicine group
Behavioral: Telemedicine — Review details of medication indication and use, activity recommendations and changes, and knowledge of arrhythmia changes and activities which are helpful with arrhythmia changes.
  Arms: Telemedicine group

SUMMARY:
The purpose of the study is to see if monthly telemedicine computer visits (visits using the computer) improve the time it takes to identify and treat an arrhythmia. The second purpose is to see if monthly telemedicine computer visits improves the participant's understanding of the arrhythmia and improves how the participant feels with daily activities.

DETAILED DESCRIPTION:
Study will utilize the Telemedicine group and the Standard Visit group (30 patients each group) to determine

Endpoints:

1. Time of recognition, time of diagnosis and time of intervention for arrhythmia. These times will be noted for each patient in each group and look for any difference in these times based upon gaining information from telemedicine visits versus 6 month follow up visit.
2. Three surveys of patient Self efficacy of medications, activity, and arrhythmia knowledge utilizing three surveys in each group. Surveys will be answered at the start of the study and end of the study by every patient within each group.

Surveys:

MUSE- Medication Understanding and Self Efficacy Tool Shortened FSES- Functioning self efficacy scale ASTA- Arrhythmia specific symptoms and health related quality of life in connection with heart rhythm disturbance

ELIGIBILITY:
Inclusion Criteria:

* Read and speak English
* 18 years of age or older
* Have a cardiac arrhythmia diagnosis
* Are willing to participate in the study and answer a pre and post survey.

Exclusion Criteria:

* Any difficulty in understanding the study
* Does not have internet or a cell phone data plan
* Any life threatening arrhythmias
* Objection to working with nurse practitioners and physician assistants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Time of recognition of an arrhythmia | Up to 6 months
  Patient recognition of a probable arrhythmia
Time of diagnosis of arrhythmia | Up to 6 months
  Time of diagnosis of arrhythmia by medical staff- at what point is the diagnosis present.
Time to treatment initiation of arrhythmia | Up to 6 months
  The time- what point in time is the treatment plan innitiated

SECONDARY OUTCOMES:
Change in self efficacy in medication use score as measured by the Medication Self Efficacy Tool (MUSE) survey | Baseline, 6 months
  MUSE is 7 items which are evaluated to identify if the patient has a good overall understanding and perception of their medicine.
Change in functioning self efficacy score as measured by the 13 Item Shortened Function Self-efficacy Scale (FSES) | Baseline, 6 months
  The FSES is 13 questions with responses scored from 1 to 5 with a maximum score of 65. Higher scores indicates higher level of functioning.
Change in self-efficacy of arrhythmia management score as measured by the Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmias (ASTA) survey | Baseline, 6 months
  The ASTA questionnaire is divided into three separate parts.
  * Part 1 is descriptive data that evaluates the patient's latest episode of arrhythmia and his/her pharmaceutical treatment.
  * Part 2 has 9 items and a four point's response scale with response alternatives from 0 to 3: "No (0), Yes, to a certain extent (1), Yes, quite a lot (2) or Yes, a lot (3) ". A summarized score is calculated for the items, a higher score implies higher symptom burden due to the heart rhythm disturbance. Scoring for the ASTA symptom burden scale ranges from 0 (least burdensome) to highest 27 (most burdensome).
  * Part 3 scale has 13 items and describes the arrhythmia's influence on daily life with a seven items physical subscale (items 1-5, 10 and 12) and a six items mental subscale (items 6-9, 11 and 13). The response alternatives from 0 to 3: "No (0), Yes, to a certain extent (1), Yes, quite a lot (2),

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Fasing, Principal Investigator — University of Michigan; Hakan Oral, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson, T, Bansler, J., Kensing, F. & Moll, J., Aligning concerns in telecare: Three concepts to guide the design of patient centered e-health, Computer supported cooperative work, 3 (6), 1181-1214, 2018.
- [Background] Dalouk K, Gandhi N, Jessel P, MacMurdy K, Zarraga IG, Lasarev M, Raitt M. Outcomes of Telemedicine Video-Conferencing Clinic Versus In-Person Clinic Follow-Up for Implantable Cardioverter-Defibrillator Recipients. Circ Arrhythm Electrophysiol. 2017 Sep;10(9):e005217. doi: 10.1161/CIRCEP.117.005217. PMID 28916510
- [Background] Dixon DL, Dunn SP, Kelly MS, McLlarky TR, Brown RE. Effectiveness of Pharmacist-Led Amiodarone Monitoring Services on Improving Adherence to Amiodarone Monitoring Recommendations: A Systematic Review. Pharmacotherapy. 2016 Feb;36(2):230-6. doi: 10.1002/phar.1697. Epub 2016 Feb 5. PMID 26846446
- [Background] Estrada JC, Darbar D. Clinical use of and future perspectives on antiarrhythmic drugs. Eur J Clin Pharmacol. 2008 Dec;64(12):1139-46. doi: 10.1007/s00228-008-0555-x. Epub 2008 Sep 2. PMID 18762931
- [Background] Goldschlager N, Epstein AE, Naccarelli GV, Olshansky B, Singh B, Collard HR, Murphy E; Practice Guidelines Sub-committee, North American Society of Pacing and Electrophysiology (HRS). A practical guide for clinicians who treat patients with amiodarone: 2007. Heart Rhythm. 2007 Sep;4(9):1250-9. doi: 10.1016/j.hrthm.2007.07.020. Epub 2007 Jul 20. PMID 17765636
- [Background] Harden M, Nystrom B, Kulich K, Carlsson J, Bengtson A, Edvardsson N. Validity and reliability of a new, short symptom rating scale in patients with persistent atrial fibrillation. Health Qual Life Outcomes. 2009 Jul 15;7:65. doi: 10.1186/1477-7525-7-65. PMID 19604399
- [Background] Honeyman, E., Ding, H., Varnfield, M., & Karunanithi, M. Mobile health applications in cardiac care. Interventional cardiology, 6.2, 227-241, 2014.
- [Background] Klein-Wiele O, Faghih M, Dreesen S, Urbien R, Abdelghafor M, Kara K, Schulte-Hermes M, Garmer M, Gronemeyer D, Hailer B. A novel cross-sector telemedical approach to detect arrhythmia in primary care patients with palpitations using a patient-activated event recorder. Cardiol J. 2016;23(4):422-8. doi: 10.5603/CJ.a2016.0033. Epub 2016 Jun 20. PMID 27320955
- [Background] Lamarche L, Tejpal A, Mangin D. Self-efficacy for medication management: a systematic review of instruments. Patient Prefer Adherence. 2018 Jul 20;12:1279-1287. doi: 10.2147/PPA.S165749. eCollection 2018. PMID 30050290
- [Background] Lowres N, Redfern J, Freedman SB, Orchard J, Bennett AA, Briffa T, Bauman A, Neubeck L. Choice of Health Options In prevention of Cardiovascular Events for people with Atrial Fibrillation (CHOICE-AF): A pilot study. Eur J Cardiovasc Nurs. 2016 Feb;15(1):39-46. doi: 10.1177/1474515114549687. Epub 2014 Sep 3. PMID 25187121
- [Background] Lopez-Villegas A, Catalan-Matamoros D, Robles-Musso E, Peiro S. Effectiveness of pacemaker tele-monitoring on quality of life, functional capacity, event detection and workload: The PONIENTE trial. Geriatr Gerontol Int. 2016 Nov;16(11):1188-1195. doi: 10.1111/ggi.12612. Epub 2015 Dec 4. PMID 26635263
- [Background] Ryan P. Integrated Theory of Health Behavior Change: background and intervention development. Clin Nurse Spec. 2009 May-Jun;23(3):161-70; quiz 171-2. doi: 10.1097/NUR.0b013e3181a42373. PMID 19395894
- [Background] Ryan P, Papanek P, Csuka ME, Brown ME, Hopkins S, Lynch S, Scheer V, Schlidt A, Yan K, Simpson P, Hoffman R; Striving to be Strong Team. Background and method of the Striving to be Strong study a RCT testing the efficacy of a m-health self-management intervention. Contemp Clin Trials. 2018 Aug;71:80-87. doi: 10.1016/j.cct.2018.06.006. Epub 2018 Jun 9. PMID 29894865
- [Background] Suter P, Suter WN, Johnston D. Theory-based telehealth and patient empowerment. Popul Health Manag. 2011 Apr;14(2):87-92. doi: 10.1089/pop.2010.0013. Epub 2011 Jan 17. PMID 21241182
- [Background] Sutton, B. D'Oranzio, Gopinethannair, R. Developing a robust monitoring program in your practice: Clinical, economic, and workflow considerations. Electrophysiology Lab Digest, 13 (2), 2013.
- [Background] Tarakji, K. For arrhythmia patients, virtual visits hold plenty of virtues. Electrophysiology consult QD, 12 (2), 2016.
- [Background] Tovel H, Carmel S. Function Self-Efficacy Scale-FSES: Development, Evaluation, and Contribution to Well-Being. Res Aging. 2016 Aug;38(6):643-64. doi: 10.1177/0164027515596583. Epub 2015 Aug 2. PMID 26239228
- [Background] Varma N, Epstein AE, Irimpen A, Schweikert R, Love C; TRUST Investigators. Efficacy and safety of automatic remote monitoring for implantable cardioverter-defibrillator follow-up: the Lumos-T Safely Reduces Routine Office Device Follow-up (TRUST) trial. Circulation. 2010 Jul 27;122(4):325-32. doi: 10.1161/CIRCULATIONAHA.110.937409. Epub 2010 Jul 12. PMID 20625110
- [Background] Varma N, Ricci RP. Telemedicine and cardiac implants: what is the benefit? Eur Heart J. 2013 Jul;34(25):1885-95. doi: 10.1093/eurheartj/ehs388. Epub 2012 Dec 4. PMID 23211231
- [Background] Walfridsson, Ulla. ASTA, University Hospital, Linkoping, Sweeden, 2012.